CLINICAL TRIAL: NCT04482348
Title: Can Crafted Communication Strategies Allow Musculoskeletal Specialists to Address Health Within the Biopsychosocial Paradigm?
Brief Title: Crafted Communication for Biopsychosocial Care in Musculoskeletal Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Professor of surgery and perioperative care, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019-01-0084
Record Dates: First submitted 2020-07-08; First posted 2020-07-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Wellness 1
Keywords: cognitive health; social health; emotional health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: New and return patients seeing an orthopedic specialist were randomized to evaluate one of 7 brief explanations of the mind-body connection with variations in cognitive, emotional, or physiology-based explanations.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- the mind is a great story teller-positively framed (Active Comparator): explanations for more pain than expected
  Interventions: Other: Explanation
- the mind is a great story teller-negatively framed (Active Comparator): explanations for more pain than expected
  Interventions: Other: Explanation
- emotionally-framed explanation-stressed or down-positive frame (Active Comparator): explanations for more pain than expected
  Interventions: Other: Explanation
- emotionally-framed explanation-stressed or down-negative frame (Active Comparator): explanations for more pain than expected
  Interventions: Other: Explanation
- mixed emotion and cognition ("mind and body work together") (Active Comparator): explanations for more pain than expected
  Interventions: Other: Explanation
- physically based explanations "over-excited state" (Active Comparator): explanations for more pain than expected
  Interventions: Other: Explanation
- physically based explanations "overstimulated" (Active Comparator): explanations for more pain than expected
  Interventions: Other: Explanation

INTERVENTIONS:
Other: Explanation — Explanation provided to patients for more pain than expected

SUMMARY:
New and return patients seeing an orthopedic specialist were randomized to evaluate one of 7 brief explanations of the mind-body connection with variations in cognitive, emotional, or physiology-based explanations. Reactions were measured as resonance (Likert scale) and Self-Assessment Manikins (SAM) for happiness, excitement, and control. Patients also completed demographic and mental and emotional health surveys. Overall 304 patients were included (mean age 49 -17, range 18 to 87; 51% men). Multilevel multivariable linear regression models were constructed to assess factors associated with resonance, happiness, excitement, and control.

DETAILED DESCRIPTION:
Study design the investigators obtained institutional review board approval and prospectively enrolled 308 patients in this cross-sectional study over a 4-month period. All patients were seen at one of four participating orthopaedic offices in a large urban area. the investigators included all new or return orthopaedic patients aged 18 to 89 years old. After the visit with the surgeon, a research assistant not involved in patient care explained the study to the patient and asked them to participate. the investigators obtained a waiver for written consent; completing the questionnaires represented consent.

Outcomes measures Each patient read one of 7 randomly selected explanations for more pain than expected on a tablet. There were 2 cognitively-framed explanations ("the mind is a great story teller"; one positively- and one negatively framed), 2 emotionally-framed explanation ("stressed or down"; one positively- and one negatively framed), one mixed emotion and cognition ("mind and body work together"), and two physically based explanations ("over-excited state", "overstimulated")

Subjects completed the following questionnaires: (1) a demographic survey including the following variables: age, sex, race/ethnicity, marital status, work status, insurance status, level of education, number of i) people living in the household, ii) children living in the household, iii) adults living in the household, iv) adults who generate income; (2) the Generalized Anxiety Disorder 2-item version (GAD-2); (3) the Patient Health Questionnaire 2-item version (PHQ-2); (4) the Pain Self-Efficacy Questionnaire 2-item version (PSEQ-2); and (5) the Pain Catastrophizing Scale 4-item version (PCS-4).

Patients rated resonance with the explanation of more pain than expected on a 5-point Likert scale as follows from 1 to 5: "nope I don't buy it", "this doesn't make sense", "I'm not sure how I feel about this", "this makes sense", and "absolutely, that makes perfect sense".

Self-Assessment Manikins (SAM; a picture-oriented instrument) were used to measure 3 affective dimensions, happiness, excitement and control in response to the explanation.

The happiness dimension ranges from a smiling happy to a frowning unhappy SAM figure. The excitement dimension ranges from an excited wide-eyed to a relaxed sleepy SAM figure. The control dimension is represented with a changing size of the SAM figure and ranges from a small to a large SAM figure; the largest represents the most control in the situation.

The GAD-2 is a 2-item questionnaire (0=not at all to 3=nearly every day) that measures symptoms of anxiety in the last two weeks. Total score ranges from 0 to 6, with higher scores indicating more symptoms of anxiety.

The PCS-4 measures less adaptive thoughts in response to nociception on a 4-item scale (0=not at all to 4=all the time). The scale contains two items on magnification, one item on rumination, and one item on helplessness. Total score ranges from 0 to 16, higher scores indicate more catastrophic thoughts.

The PSEQ-2 measures two beliefs: that one can engage in activities and enjoy life in spite of pain. The total score ranges from 0 (not at all confident) to 12 (completely confident).

The PHQ-2 is a 2-item questionnaire that measures symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* all new or return orthopaedic patients aged 18 to 89 years old

Exclusion Criteria:

* Illiteracy
* Cognitive problems which patient was not able to fill surveys

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
resonance with the explanation of more pain than expected | up to 24 weeks
  Patients rated resonance with the explanation of more pain than expected on a 5-point Likert scale from 1 to 5, as follows: "nope, I don't buy it," "this doesn't make sense," "I'm not sure how I feel about this," "this makes sense," and "absolutely, that makes perfect sense." Likert scales are valid for measuring variation in opinion. This specific Likert scale is new and specific to this study, and so no minimum clinically important difference has been defined. Given how the scale is anchored, a difference of about 1 point seems relevant.
Self-Assessment Manikins(SAM) | up to 24 weeks
  Self-assessment manikins (SAMs), a picture-oriented instrument, were used to measure three affective dimensions of happiness, stimulation/excitement, and security/control in response to the explanations. The happiness dimension ranges from a smiling, happy SAM figure to a frowning, unhappy figure. The excitement dimension ranges from an excited, wide-eyed SAM figure to a relaxed, sleepy figure. The control dimension is represented by an SAM figure that changes in size and ranges from a small SAM figure to a large one; the largest figure represents the greatest feeling of security and control. With respect to written explanations of the mind-body connection, we favored greater feelings of happiness and control and relatively neutral feelings of excitement.

SECONDARY OUTCOMES:
demographic survey | up to 24 weeks
  age, sex, race/ethnicity, marital status, work status, insurance status, level of education, number of i) people living in the household, ii) children living in the household, iii) adults living in the household, iv) adults who generate income
GAD-2 | up to 24 weeks
  a 2-item questionnaire (0=not at all to 3=nearly every day) that measures symptoms of anxiety in the last two weeks. Total score ranges from 0 to 6, with higher scores indicating more symptoms of anxiety
PCS-4 | up to 24 weeks
  measures less adaptive thoughts in response to nociception on a 4-item scale (0=not at all to 4=all the time). The scale contains two items on magnification, one item on rumination, and one item on helplessness. Total score ranges from 0 to 16, higher scores indicate more catastrophic thoughts
PSEQ-2 | up to 24 weeks
  measures two beliefs: that one can engage in activities and enjoy life in spite of pain. The total score ranges from 0 (not at all confident) to 12 (completely confident).
PHQ-2 | up to 24 weeks
  a 2-item questionnaire (0=not at all to 3=nearly every day) that measures symptoms of depression in the last two weeks. Total score ranges from 0 to 6, with higher scores indicating more symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Dell Medical School, University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez AI, Kortlever JTP, Brown LE, Ring D, Queralt M. Can Crafted Communication Strategies Allow Musculoskeletal Specialists to Address Health Within the Biopsychosocial Paradigm? Clin Orthop Relat Res. 2021 Jun 1;479(6):1217-1223. doi: 10.1097/CORR.0000000000001635. PMID 33411452